CLINICAL TRIAL: NCT02500173
Title: Analysis of Effects and Side Effects in Patients Undergoing Radiation Therapy - Quality Control Using Clinical Database
Brief Title: Analysis of Effects and Side Effects in Patients Undergoing Radiation Therapy
Status: Terminated | Type: Observational
Why Stopped: General Informed Consent has been introduced at the Hospital, no need for study anymore
Sponsor: Kantonsspital Graubuenden (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr.2015-0221
Record Dates: First submitted 2015-06-18; First posted 2015-07-16 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Cancer
Keywords: radiotherapy; side effects
MeSH Terms: conditions — Neoplasms | interventions — Radiation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Radiation — Radiation therapy

SUMMARY:
To collect and analyze effects and side effects in patients undergoing radiotherapy.

This study investigates how analysis of effects and side effects will influence outcome of patients. These retrospectively collected data allow to adapt and improve radiotherapy treatment regimens .

DETAILED DESCRIPTION:
Effects and side effects in patients undergoing radiotherapy will be collected over the next five years (2015-2020). It is planned to include 600 to 650 new patients referred for radiotherapy per calender year. It is estimated that 3000 patients will be included at the end of the study after five years. Patient Information on diseae and treatment will be collected and analyzed. Common statistical algorithms will be performed for outcome analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing radiotherapy at the Kantonsspital Graubuenden

Exclusion Criteria:

* No radiotherapy at Kantonsspital Graubuenden
* Age: < 20 years, > 105 years

Ages: 20 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing radiotherapy at the Kantonsspital Graubuenden
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Side effects in patients undergoing radiotherapy (CTCAE v4.03) | 5 Years
  acute and late side effects according to CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Zwahlen, MD MBA, Study Chair — Kantonsspital Winterthur, Department of Radiation Oncology
Locations (1):
- Kantonsspital Graubuenden, Department of Radiaton Oncology, Chur, Switzerland

IPD SHARING:
Plan to Share IPD: No